CLINICAL TRIAL: NCT05495880
Title: Forearm-Supported Head Extension to Decrease Dental Contact Between Laryngoscope Blade and Maxillary Incisors During Direct Laryngoscopy
Brief Title: Forearm-Supported Head Extension to Decrease Dental Contact
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_novel_intu
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-08

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forearm-supported (Experimental): forearm-supported head extension during direct laryngoscopy
  Interventions: Procedure: Laryngoscopy with forearm-support
- Control (Active Comparator): without forearm-support for head extension during direct laryngoscopy
  Interventions: Procedure: Laryngoscopy without forearm-support

INTERVENTIONS:
Procedure: Laryngoscopy with forearm-support — forearm-supported head extension during direct laryngoscopy
  Arms: Forearm-supported
Procedure: Laryngoscopy without forearm-support — without forearm-support for head extension during direct laryngoscopy
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether the forearm-supported head extension decreases dental contact between laryngoscope blade and maxillary incisors during direct laryngoscopy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery that require endotracheal intubation for general anesthesia

Exclusion Criteria:

* Trauma or disease or cervical spine
* Toothless patient
* Dentoalveolar injury
* Anatomical anomaly of face or airway
* History of difficult intubation
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-05-18 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dental contact | during laryngoscopy
  Dental contact between laryngoscope blade and maxillary incisors (Y/N)

SECONDARY OUTCOMES:
Blade-to-tooth distance | during laryngoscopy
  Teeth distance between laryngoscope blade and maxillary incisors (mm)
Angle of head extension | during laryngoscopy
  Angle of head extension during direct laryngoscopy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song SE, Ju JW, Park JY, Park D, Yoon S, Nam K, Lee HJ, Seo JH, Kim WH, Bahk JH. Forearm support to reduce dental contact during direct laryngoscopy: a randomized crossover trial. Can J Anaesth. 2025 Oct;72(10):1511-1520. doi: 10.1007/s12630-025-03035-w. Epub 2025 Oct 13. PMID 41083757